CLINICAL TRIAL: NCT02796456
Title: Determination of Maternal and Neonatal Apelinemia in Obese Women During Pregnancy
Acronym: OB-APE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014_70; 2015-A01696-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-05-19; First posted 2016-06-10 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Pregnancy; Gestational Diabetes
Keywords: apelin; colostrum; plasma; glycemic markers; lipidic markers; pregnancy; postpartum
MeSH Terms: conditions — Obesity; Diabetes, Gestational | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Placenta samples will be collected and RT-qPCR will be done to analyze RNA in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal weight women: BMI between 18.5 and 25 kg/m2 and without gestational diabetes
  Interventions: Other: blood sample
- Obese women without gestational diabetes: BMI more than 30 kg/m2 and without gestational diabetes
  Interventions: Other: blood sample
- Obese women with gestational diabetes: BMI more than 30 kg/m2 and with gestational diabetes
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
Background :

Apelin and its receptor APJ have been implicated in pathologies including cardiovascular disease, diabetes and obesity. Little is known about the function of the apelinergic system during gestation.

Objective :

The main objective of this study is to compare apelinemia in fasting normal weight and obese women at the end of pregnancy, between 35 and 41 weeks of gestation (WG).

Strategy and method:

A prospective research evaluating will be conducted to compare apelinemia in fasting normal weight and obese women at the end of pregnancy, between 35 and 41 weeks of gestation (WG).

A third group will be created to check if gestational diabetes is not a confounding factor in obesity (group of obese women with gestational diabetes).

Investigators will try to see if apelinemia is correlated to lipidic and glycemic markers.

Samples will be collected in the cord blood to compare maternal and neonatal apelinemia and to see if neonatal apelinemia is correlated to the child's weight and birth size and to the weight of the placenta.

Placenta samples will be collected and RT-qPCR will be done to analyze RNA in each group.

Two days after delivery, obese and not obese women will be fasted and plasma and colostrum will be collected. Investigators will compare apelin levels in the colostrum between these 2 groups and then investigators will try to see if apelin level is correlated in the colostrum and in maternal plasma.

DETAILED DESCRIPTION:
Background :

Apelin and its receptor APJ have been implicated in pathologies including cardiovascular disease, diabetes and obesity.

Little is known about the function of the apelinergic system during gestation.

In a previous study, investigators evaluated in mice this system at the feto-maternal interface in insulin-resistant obese female (HF) mice. Maternal apelinemia was decreased at term and fetal apelinemia was sixfold higher than maternal level. Ex-vivo, the placenta releases high amount of apelin at E12.5 and E18.5. In HF pregnant mice at term, apelinemia as well as placental apelin and APJ mRNA levels were increased whereas placental release of apelin was drastically reduced.

ELIGIBILITY:
Inclusion Criteria:

* Obese pregnant women
* Age from 18 to 42 years old
* Singleton pregnancy between 35+0 to 41+6 weeks of pregnancy

Exclusion Criteria:

* Severe heart, liver or kidney disease
* Multiple pregnancy
* Hypertension, preeclampsia, small for gestational age
* Pre-gestational diabetes
* Bariatric surgery
* Medication other than normal pregnancy supplementations
* Tabacco or drugs consummation during pregnancy
* Provided artificial feeding
* Fetal anoxia with cord pH less than 7.0
* Genetic or chromosomal mother's and / or newborn's abnormality
* Fetal malformation
* Trusteeship or tutorship
* Refusal to participate in research
* Unable to attend the entire study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between 18 and 42 years old, pregnant, between 35 and 40 WG.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Biological measure : Maternal apelinemia (Plasma Concentration) | between 35 and 41 weeks of gestation (WG)
  plasma sample

SECONDARY OUTCOMES:
Biological measure : Neonatal apelinemia (Plasma Concentration) | the day of the delivery
  plasma sample
Biological measure : Maternal apelinemia (Plasma Concentration) | the day of the delivery and 2 days after the delivery
  plasma sample
apelin level in the colostrum | 2 days after the delivery
  colostrum sample
C-peptide | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
glycemia | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
insulinemia | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
C-peptide | the day of the delivery
  neonatal plasma sample
glycemia | the day of the delivery
  neonatal plasma sample
insulinemia | the day of the delivery
  neonatal plasma sample
total cholesterol | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
HDL | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
LDL | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
triglycerides | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
apolipoprotein A | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
apolipoprotein B | between 35 and 41 weeks of gestation (WG) and 2 days after the delivery
  maternal plasma sample
total cholesterol | the day of the delivery
  neonatal plasma sample
Biological measure : HDL | the day of the delivery
  neonatal plasma sample
Biological measure : LDL | the day of the delivery
  neonatal plasma sample
triglycerides | the day of the delivery
  neonatal plasma sample
apolipoprotein A | the day of the delivery
  neonatal plasma sample
apolipoprotein B | the day of the delivery
  neonatal plasma sample
BMI | at baseline
  measure maternal gain of weight before pregnancy and during pregnancy in maternal declaration
Infant weight | within 2 days of postpartum
Infant size | within 5 days of postpartum
Placenta weight | the days of the delivery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Deruelle, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandre - CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided